CLINICAL TRIAL: NCT03164200
Title: An Egg Based Breakfast Maintains Flexibility in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Barbara Gower, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2148
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Diabetes; Heart Diseases
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases

STUDY DESIGN:
Masking Description: Patients were randomized to either a egg breakfast or a carbohydrate breakfast
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fat breakfast (Experimental): 45% fat 35% Carbohydrate 20% protein
  Interventions: Other: High fat breakfast
- Higher carbohydrate breakfast (Experimental): 60% carbohydrate 20% fat 20% protein
  Interventions: Other: Higher carbohydrate breakfast

INTERVENTIONS:
Other: High fat breakfast — High fat breakfast
  Arms: High fat breakfast
Other: Higher carbohydrate breakfast — Higher carbohydrate breakfast
  Arms: Higher carbohydrate breakfast

SUMMARY:
Aging is associated with an increased risk for metabolic diseases, such as type 2 diabetes and cardiovascular disease. There is reason to believe that the time of day when specific food groups are eaten affects this risk. The investigators propose that eating foods made up of fat and protein (such as eggs) in the morning for breakfast, rather than foods made up of carbohydrates (such as white-bread toast or sugary cereal) may promote a healthier metabolism. This is because the body is designed to burn fat during times of fasting, such as overnight, during sleep. Thus, the body is not prepared to burn sugar early in the morning, when most people eat breakfast. Studies with mice have shown that a sugary breakfast meal inhibits the ability of the body to burn fat for the entire day. In contrast, a breakfast meal with more fat enabled the animals to burn fat as well as other fuels throughout the day. The ability to burn fat is thought to minimize risk for obesity, as well as related diseases such as type 2 diabetes and heart disease. The purpose of this study is to determine if, in older adult humans, consumption of a lower-carbohydrate breakfast meal (relative to a higher-carbohydrate meal) is associated with a healthier metabolism.

ELIGIBILITY:
Inclusion Criteria:

* • Age 55-75

  * Body mass index 24-29 kg/m2

Exclusion Criteria:

* • Current practice of greater than 2h/wk of moderate intentional exercise

  * Uncontrolled diabetes
  * Unwillingness to eat study diets
  * Use of any medication known to affect metabolism
  * History of eating disorder
  * Difficulty chewing and swallowing solid food
  * Digestive diseases
  * Cognitive impairment
  * Depression
  * Recent weight change (+/- 10 lbs. in the last 12 mo.)
  * Poorly controlled blood pressure (SBP > 159 or DBP >95 mm Hg)
  * History of non-skin cancer in the last 5 y
  * Cardiovascular disease event in the past 6 mo.
  * Severe pulmonary disease
  * Renal failure
  * Major liver dysfunction (elevation of liver transaminases >3x normal in past 2 y; current/recent smoker (within 6 mo.)
  * Use of estrogen or testosterone replacement therapy
  * Current use of oral corticosteroids >5 days/month on average
  * Current use of medications for treatment of psychosis or manic-depressive illness
  * Use of weight loss medications in the previous 3 months
  * Unable to adhere to diet recommendations

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2013-10-30 (Actual); Study Completion 2013-10-30 (Actual)

PRIMARY OUTCOMES:
Respiratory quotient (RQ, a measure of substrate oxidation) | 4 weeks
  24 hour respiratory quotient will be measured using whole-room indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gower, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bush NC, Resuehr HES, Goree LL, Locher JL, Bray MS, Soleymani T, Gower BA. A High-Fat Compared with a High-Carbohydrate Breakfast Enhances 24-Hour Fat Oxidation in Older Adults. J Nutr. 2018 Feb 1;148(2):220-226. doi: 10.1093/jn/nxx040. PMID 29490097